CLINICAL TRIAL: NCT01143701
Title: Evaluation of an Intervention for Improving Community-based Pediatric ADHD Care
Brief Title: Evaluation of an Intervention for Improving Community-based Pediatric Attention-Deficit Hyperactivity Disorder (ADHD) Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nationwide Children's Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeff Epstein, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MH083665; 1R01MH083665-01A2 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADHD Collaborative Intervention (Experimental): The ADHD Collaborative intervention model includes academic detailing, quality improvement methods, and innovative tools (e.g., web portal) designed to promote and support the systematic use of the American Academy of Pediatrics consensus recommendation for evidence-based ADHD care.
  Interventions: Other: ADHD Collaborative
- Typical ADHD care (No Intervention): Physicians in this group will provide typical ADHD care.

INTERVENTIONS:
Other: ADHD Collaborative — The ADHD Collaborative intervention model includes academic detailing, quality improvement methods, and innovative tools (e.g., web portal) designed to promote and support the systematic use of the AAP guidelines.
  Arms: ADHD Collaborative Intervention

SUMMARY:
ADHD is the most prevalent mental health disorder of childhood. The majority of children with ADHD receive their care in primary care settings. While the American Academy of Pediatrics (AAP) issued evidence-based guidelines and recommendations for pediatricians, most pediatricians have difficulty adhering to these guidelines. Given observed deficiencies in evidence-based ADHD care and the likely effects on child outcomes, the development and testing of interventions aimed at improving ADHD care in primary care settings is necessary. Cincinnati Children's Hospital Medical Center has developed a model intervention, termed the ADHD Collaborative, to comprehensively address this issue. The ADHD Collaborative intervention model includes academic detailing, quality improvement methods, and innovative tools (e.g., web portal) designed to promote and support the systematic use of the AAP guidelines. This intervention model has been used to train over 200 physicians at 55 practices in the Greater Cincinnati area. The intervention appears to produce 2- to 4-fold increases in the use of evidence-based ADHD-related practice behaviors in participating physicians. To date, the intervention has been implemented as a quality improvement project with few experimental controls. The primary goal of the proposed study is to conduct an experimentally-controlled cluster randomized trial of the ADHD Collaborative intervention. Thirty-two pediatric practices will be randomly assigned to receive the ADHD Collaborative intervention or to provide usual care. Approximately 96 physicians and 576 of their ADHD patients will be included in the study. Chart reviews, parental interviews, and parent and teacher rating scales will be collected. Between- and within-group hierarchical linear modeling analyses will examine whether the intervention produces significant improvements in pediatrician practice behaviors, patient satisfaction with ADHD care, and child outcomes over and above typical ADHD care. Also, the relative cost effectiveness of the ADHD Collaborative intervention over typical care will be established by computing incremental cost-effectiveness ratios using cost and effect size estimates.

ELIGIBILITY:
Inclusion Criteria:

* Practice must have a minimum of two pediatricians who agree to participate.
* Practice must have an electronic billing system.
* Practice must have internet access at office.
* Practice must not have an on-site mental health professional.
* Practice must have a member of practice staff willing to be trained in human subjects certification and willing to consent families.
* Children must be in Grade 1-5.
* Children must be newly diagnosed with ADHD.

Exclusion Criteria:

-

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 577 (Actual)
Dates: Start 2010-05; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Childrens Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Gordon MK, Baum RA, Gardner W, Kelleher KJ, Langberg JM, Brinkman WB, Epstein JN. Comparison of Performance on ADHD Quality of Care Indicators: Practitioner Self-Report Versus Chart Review. J Atten Disord. 2020 Aug;24(10):1457-1461. doi: 10.1177/1087054715624227. Epub 2016 Jan 28. PMID 26823383
- [Background] Brinkman WB, Baum R, Kelleher KJ, Peugh J, Gardner W, Lichtenstein P, Langberg J, Epstein JN. Relationship Between Attention-Deficit/Hyperactivity Disorder Care and Medication Continuity. J Am Acad Child Adolesc Psychiatry. 2016 Apr;55(4):289-94. doi: 10.1016/j.jaac.2016.02.001. Epub 2016 Feb 5. PMID 27015719
- [Background] Epstein JN, Kelleher KJ, Baum R, Brinkman WB, Peugh J, Gardner W, Lichtenstein P, Langberg J. Variability in ADHD care in community-based pediatrics. Pediatrics. 2014 Dec;134(6):1136-43. doi: 10.1542/peds.2014-1500. Epub 2014 Nov 3. PMID 25367532
- [Background] Epstein JN, Langberg JM, Lichtenstein PK, Kolb R, Simon JO. The myADHDportal.com Improvement Program: An innovative quality improvement intervention for improving the quality of ADHD care among community-based pediatricians. Clin Pract Pediatr Psychol. 2013 Mar 1;1(1):55-67. doi: 10.1037/cpp0000004. PMID 24163788
- [Result] Epstein JN, Kelleher KJ, Baum R, Brinkman WB, Peugh J, Gardner W, Lichtenstein P, Langberg JM. Impact of a Web-Portal Intervention on Community ADHD Care and Outcomes. Pediatrics. 2016 Aug;138(2):e20154240. doi: 10.1542/peds.2015-4240. PMID 27462065

RESULTS

PARTICIPANT FLOW:
Groups:
- ADHD Collaborative Intervention: The ADHD Collaborative intervention model includes academic detailing, quality improvement methods, and innovative tools (e.g., web portal) designed to promote and support the systematic use of the American Academy of Pediatrics consensus recommendation for evidence-based ADHD care.
  ADHD Collaborative: The ADHD Collaborative intervention model includes academic detailing, quality improvement methods, and innovative tools (e.g., web portal) designed to promote and support the systematic use of the American Academy of Pediatrics ADHD guidelines.
Period: Overall Study
Arm/Group | ADHD Collaborative Intervention | Typical ADHD Care
Started | 258 | 319
Completed | 235 (Number of patients for whom at least one set of post-baseline parent-ratings were collected) | 287 (Number of patients for whom at least one set of post-baseline parent-ratings were collected)
Not Completed | 23 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADHD Collaborative Intervention | Typical ADHD Care | Total
Number analyzed (Participants) | 258 | 319 | 577
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.9 (1.5) | 7.8 (1.4) | 7.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 91 | 170
  Male | 179 | 228 | 407
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 252 | 312 | 564
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 90 | 123
  White | 187 | 191 | 378
  More than one race | 36 | 35 | 71
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 258 | 319 | 577

OUTCOME MEASURES:

1. Primary Outcome: Parent-rated ADHD Symptoms
Description: Total Symptom Score on Parent-Rated Vanderbilt ADHD Rating Scale (range=0-54). Higher scores represent more severe ADHD symptom presentation.
Time Frame: 12 months
Population: Hierarchical Modeling accounted for clustering of patients nested within providers and providers nested within practices.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Practices Analyzed
Arm/Group | ADHD Collaborative Intervention | Typical ADHD Care
Number analyzed (Participants) | 235 | 287
Number analyzed (Practices Analyzed) | 22 | 22
scores on a scale | 20.5 (9.0) | 24.1 (9.4)
Statistical Analysis 1: Comparison: ADHD Collaborative Intervention vs Typical ADHD Care; Utilizing the full sample (n=577), an intent-to-treat analyses was conducted comparing patient outcomes across intervention and control groups using a three-level mixed model. Baseline ratings were entered as a covariate. Post-baseline ratings collected closest to 12-months post-baseline were entered as dependent variables; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-5.89 to -1.19]

2. Primary Outcome: Teacher-rated ADHD Symptoms
Description: Total Symptom Score on Teacher-Rated Vanderbilt ADHD Rating Scale (range=0-54). Higher scores represent more severe ADHD symptom presentation.
Time Frame: 12 months
Population: Analyses only included patients who had a post-intervention teacher-rated ADHD scale. Hierarchical Modeling accounted for clustering of patients nested within providers and providers nested within practices.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Practices Analyzed
Arm/Group | ADHD Collaborative Intervention | Typical ADHD Care
Number analyzed (Participants) | 132 | 164
Number analyzed (Practices Analyzed) | 22 | 22
scores on a scale | 19.0 (9.9) | 20.4 (11.1)
Statistical Analysis 1: Comparison: ADHD Collaborative Intervention vs Typical ADHD Care; An intent-to-treat analyses was conducted comparing patient outcomes across intervention and control groups using a three-level mixed model. Baseline ratings were entered as a covariate. Post-baseline ratings collected closest to 12-months post-baseline were entered as dependent variables; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-4.71 to 1.75]

ADVERSE EVENTS:
Arm/Group | ADHD Collaborative Intervention | Typical ADHD Care
Serious Adverse Events (participants affected / at risk) | 0/258 | 0/319
Other Adverse Events (participants affected / at risk) | 0/258 | 0/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No